CLINICAL TRIAL: NCT06188299
Title: The Effects Of Intraoperative Different Fluid Therapy Protocols On Postoperative Renal Functions
Brief Title: Intraoperative Different Fluid Therapy Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2-21-1078
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Intraoperative Fluid Management
Keywords: Liberal Fluid Therapy; Restrictive Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Liberal Fluid Therapy Group and Targeted Fluid Therapy Groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Group Therapy (No Intervention): Liberal Fluid Therapy was administered to this group. Fluid restrictions were not used.
- Targeted Fluid Therapy (Other): Targeted (restrictive) Fluid therapy was administered to this group. Fluids were given according to targeted blood pressure levels and aimed to avoid from fluid overload.
  Interventions: Other: Restricted Fluid Administration

INTERVENTIONS:
Other: Restricted Fluid Administration — Restrictive fluid administration generally consists of partial or no replacement for the intravascular expansion from anesthesia, in which case vasopressors are usually administered, no replacement for the third space loss, and only partial replacement for deficits from preoperative fasting.
  Arms: Targeted Fluid Therapy

SUMMARY:
We aimed to evaluate the relationship between different intraoperative fluid therapy protocols and postoperative renal damage and mortality.

DETAILED DESCRIPTION:
Sixty patients who 18-65 age and underwent pancreatic surgery in our hospital were included in the study. They were divided into two groups as liberal fluid therapy (Group 1, n=30) and targeted fluid therapy (Group 2, n=30).

ELIGIBILITY:
Inclusion Criteria:

* Planned pancreatic surgery

Exclusion Criteria:

* No exclusion criteria was presetted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
AKI | 72 Hour
  Postoperative Renal Injury
Mortality | 72 Hour
  Intraoperative and Postoperative Mortality Rate

SECONDARY OUTCOMES:
Blood Loss | Intraoperative period
  Intraoperative total blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messina A, Robba C, Calabro L, Zambelli D, Iannuzzi F, Molinari E, Scarano S, Battaglini D, Baggiani M, De Mattei G, Saderi L, Sotgiu G, Pelosi P, Cecconi M. Association between perioperative fluid administration and postoperative outcomes: a 20-year systematic review and a meta-analysis of randomized goal-directed trials in major visceral/noncardiac surgery. Crit Care. 2021 Feb 1;25(1):43. doi: 10.1186/s13054-021-03464-1. PMID 33522953
- [Background] Oh TK, Song IA, Do SH, Jheon S, Lim C. Association of perioperative weight-based fluid balance with 30-day mortality and acute kidney injury among patients in the surgical intensive care unit. J Anesth. 2019 Jun;33(3):354-363. doi: 10.1007/s00540-019-02630-8. Epub 2019 Mar 27. PMID 30919134
- [Background] Bihari S, Dixon DL, Painter T, Myles P, Bersten AD. Understanding Restrictive Versus Liberal Fluid Therapy for Major Abdominal Surgery Trial Results: Did Liberal Fluids Associate With Increased Endothelial Injury Markers? Crit Care Explor. 2021 Jan 25;3(1):e0316. doi: 10.1097/CCE.0000000000000316. eCollection 2021 Jan. PMID 33521643
- [Background] Mason SA, Nathens AB, Finnerty CC, Gamelli RL, Gibran NS, Arnoldo BD, Tompkins RG, Herndon DN, Jeschke MG; Inflammation and the Host Response to Injury Collaborative Research Program.. Hold the Pendulum: Rates of Acute Kidney Injury are Increased in Patients Who Receive Resuscitation Volumes Less than Predicted by the Parkland Equation. Ann Surg. 2016 Dec;264(6):1142-1147. doi: 10.1097/SLA.0000000000001615. PMID 27828823
- [Background] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Background] Gottin L, Martini A, Menestrina N, Schweiger V, Malleo G, Donadello K, Polati E. Perioperative Fluid Administration in Pancreatic Surgery: a Comparison of Three Regimens. J Gastrointest Surg. 2020 Mar;24(3):569-577. doi: 10.1007/s11605-019-04166-4. Epub 2019 Apr 3. PMID 30945088
- [Background] Yilmaz G, Akca A, Kiyak H, Can E, Aydin A, Salihoglu Z. Pleth Variability Index-Based Goal-Directed Fluid Management in Patients Undergoing Elective Gynecologic Surgery. Sisli Etfal Hastan Tip Bul. 2022 Jun 28;56(2):220-226. doi: 10.14744/SEMB.2021.81073. eCollection 2022. PMID 35990294
- [Background] Collange O, Jazaerli L, Lejay A, Biermann C, Caillard S, Moulin B, Chakfe N, Severac F, Schaeffer M, Mertes PM, Steib A. Intraoperative Pleth Variability Index Is Linked to Delayed Graft Function After Kidney Transplantation. Transplant Proc. 2016 Oct;48(8):2615-2621. doi: 10.1016/j.transproceed.2016.06.046. PMID 27788791
- [Background] Demirel I, Bolat E, Altun AY, Ozdemir M, Bestas A. Efficacy of Goal-Directed Fluid Therapy via Pleth Variability Index During Laparoscopic Roux-en-Y Gastric Bypass Surgery in Morbidly Obese Patients. Obes Surg. 2018 Feb;28(2):358-363. doi: 10.1007/s11695-017-2840-1. PMID 28762023
- [Background] Fischer MO, Lemoine S, Tavernier B, Bouchakour CE, Colas V, Houard M, Greub W, Daccache G, Hulet C, Compere V, Taing D, Lorne E, Parienti JJ, Hanouz JL; Optimization using the Pleth Variability Index (OPVI) Trial Group. Individualized Fluid Management Using the Pleth Variability Index: A Randomized Clinical Trial. Anesthesiology. 2020 Jul;133(1):31-40. doi: 10.1097/ALN.0000000000003260. PMID 32205547